CLINICAL TRIAL: NCT01131650
Title: Prevalence of Diabetic Retinopathy in São José do Rio Preto-SP-Brazil
Status: Completed | Type: Observational
Sponsor: Hospital do Olho Rio Preto (Other)
Collaborators: Faculty of Medicine of Ribeirão Preto (FMRP-USP) (Other)
Responsible Party: CARLOS EDUARDO CURY JUNIOR
Other Study IDs: mc201106
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Diabetic Retinopathy
Keywords: Prevalence of diabetic retinopathy; Diabetes; Retinopathy; Prevalence; Population
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus; Retinal Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- diabetic retinopathy
- diabetica retinopathy prevalence

SUMMARY:
Prevalence of Diabetic Retinopathy in São José do Rio Preto-SP-Brazil

Abstract

Objective: To determine the prevalence and characteristics of diabetic retinopathy (DR) among patients from São José do Rio Preto-SP-Brazil .

Local: Departamento de Retina e Vítreo do Hospital do Olho de Rio Preto (HORP)

Methods: Design: population-based cross-sectional study. The study sample, of 710 patients was derived from the HIPERDIA (Diabetes and High-blood pressure social health care program) of São José do Rio Preto . All patients , known to have diabetes , underwent an eye examination by biomicroscope and indirect ophthalmoscope to check for any signs of DR through dilated pupils. Participants were also interviewed and examined to determine their demographic characteristics, medical conditions and the realization of previous fundoscopic eye examination. Statistical studies were done with t -Student test , Fisher test or chi-square test.

DETAILED DESCRIPTION:
Prevalence of Diabetic Retinopathy in São José do Rio Preto-SP-Brazil

Abstract

Objective: To determine the prevalence and characteristics of diabetic retinopathy (DR) among patients from São José do Rio Preto-SP-Brazil .

Local: Departamento de Retina e Vítreo do Hospital do Olho de Rio Preto (HORP)

Methods: Design: population-based cross-sectional study. The study sample, of 710 patients was derived from the HIPERDIA (Diabetes and High-blood pressure social health care program) of São José do Rio Preto . All patients , known to have diabetes , underwent an eye examination by biomicroscope and indirect ophthalmoscope to check for any signs of DR through dilated pupils. Participants were also interviewed and examined to determine their demographic characteristics, medical conditions and the realization of previous fundoscopic eye examination. Statistical studies were done with t -Student test , Fisher test or chi-square test.

Results: Among 710 screened patients 112 had some degree of diabetic retinopathy and the overall standardized prevalence of any retinopathy was 16,3%., including 90 (80,4%) with non-proliferative and (22) 19,6 % with proliferative diabetic retinopathy. Only 143 patients (68,7%) had a history of previous fundoscopic eye examination.

Conclusion: This study demonstrated that DM and their complications are a important public health problem. The duration of DM and glicemic control is strongly associated with DR . Prevention programs with periodic fundoscopic exams shows to diminished the prevalence of this ocular disease.

Keywords: Diabetes, Retinopathy, Prevalence, Population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Diabetes Melittus

Exclusion Criteria:

* Patients without Diabetes Melittus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study sample, of 710 patients was derived from the HIPERDIA (Diabetes and High-blood pressure social health care program) of São José do Rio Preto
Sampling Method: Probability Sample
Enrollment: 710 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of diabetic retinopathy

SECONDARY OUTCOMES:
associated risk factors of diabetic retinopathy

CONTACTS AND LOCATIONS:
Locations (1):
- Carlos Eduardo Cury Junior, São José do Rio Preto, São Paulo, Brazil